CLINICAL TRIAL: NCT03644914
Title: Enhancing Reading Skills in 1st Grade Children Identified as Reading Below Grade Level
Brief Title: Enhancing Reading Skills in 1st Grade Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Sharon Gutman, Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAR8813
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Literacy
Keywords: Reading; 1st grade; Literacy
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Intervention Model Description: Intervention will take place in a New York City (NYC) elementary school. 24 first graders, identified by their teachers as reading below grade level, will be randomized to an intervention or control group. The 12 participants randomized to the intervention group will receive the 10-week reading program, twice weekly in 1-hour sessions. The Co-I and child will work together in individual sessions on sight recognition and phonetic decoding of words established as meeting 1st grade essential literacy standards. Intervention will incorporate word recognition and phonetic decoding within the context of games and play in which the child is able to move about and associate words with color, video, and music. Intervention will also use each child's personal interests as a context around which sight words will be learned. Control group participants will not receive intervention. Both the intervention and control group participants will continue to receive typical classroom reading instruction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Reading Program) (Experimental): First graders who will receive the 10-week reading program (a total of 20 hours), twice weekly in 1-hour sessions, and will continue to receive typical classroom reading instruction.
  Interventions: Behavioral: 10-week Reading Program
- Control Group (No Intervention): First graders who will not take part in the reading program but will continue to receive typical classroom reading instruction.

INTERVENTIONS:
Behavioral: 10-week Reading Program — Intervention sessions will be carried out during the school day in a private school room. In each session, the investigator will work with the child individually to help him or her read better. Intervention will incorporate word recognition and phonetic decoding of words established as meeting 1st grade essential literacy standards. Learning techniques will involve games, play, movement, music, and breaks (i.e., the child is able to move about and associate words with color, video, and music. Three 5-minute breaks will be integrated into each 1-hour session to allow the child time to rest and process learned material). Intervention will also use each child's personal interests as a context around which sight words will be learned.
  Arms: Intervention Group (Reading Program)

SUMMARY:
The purpose of the present study is to assess a reading intervention for first graders who are identified by their teachers as reading below grade level. The intervention addresses reading skills through a variety of techniques including games, play, movement exercises, music, and breaks to enhance literacy skills and reduce frustration commonly accompanying sight word recognition and phonemic decoding.

Over half of elementary school students in the United States are reading below grade level compared to their same age peers. Children with poor reading skills are more likely to experience academic and behavioral problems. When students are not reading at grade level by 4th grade, they are more likely to experience future academic failure, school dropout, juvenile delinquency, teenage pregnancy, and under- or unemployment in adulthood. Traditional methods of classroom large group instruction require children to sit quietly and concentrate on small print for extended periods of time. Many children experience frustration and agitation in response to such reading demands.

DETAILED DESCRIPTION:
The National Assessment of Educational Progress estimates that only 35% of fourth graders in the United States are able to read at or above grade level. Children's future academic success is accurately predicted by performance in the first three years of school. A student is four times more likely to drop out of high school if he or she is not reading proficiently by the end of third grade. High school dropouts are three times more likely to be unemployed than college graduates per US Bureau of Labor Statistics in 2018, and those who are employed earn an average of 61% less over the course of their lifetimes compared to their college-educated peers per US Census Bureau in 2012. Eighty-five percent of juveniles facing trial in the court system are functionally illiterate per National Criminal Justice Reference Service in 2003, and adolescent girls with low literacy skills are five times more likely to become pregnant than teenagers who can read at or above grade level.

Despite the preponderance of data expounding a literacy crisis in the US, the status quo of reading instruction in US elementary schools has not been effective in remediating functional illiteracy. In classrooms averaging 21.6 students, teachers are unable to provide the individualized instruction that is necessary to meet the learning needs of at-risk students. Reading specialists who work with children one-on-one and in small groups employ methods similar to those of classroom teachers, requiring children to sit quietly and sustain their attention on small print. These demands are difficult for children experiencing challenges with self-regulation, and school environments requiring these behaviors for several hours each day may inculcate feelings of frustration and failure in the children who most need to develop a sense of self-efficacy as readers with full membership in the world of print. In this study, twenty-four first graders will be assigned by chance to a reading or no-reading group.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a NYC elementary school in 1st grade
* Between 6-7 years old
* Identified by teachers as reading below 1st grade level

Exclusion Criteria:

* Children with severe behavioral problems making cooperation with intervention procedures difficult

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Test of Word Reading Efficiency (TOWRE) Score | Post-intervention (10 weeks)
  The TOWRE is a measure of reading fluency and accuracy for both children and adults. The instrument consists of two subtests: sight word efficiency (108 word items) and phonemic decoding efficiency (66 word items). The subtests can be scored separately or aggregately for a total score. Scores are calculated based on the number of total words read correctly in a 45 second period. Administration requires approximately 10 minutes.

SECONDARY OUTCOMES:
Change in Inventory of Reading Occupations (IRO) Score | Post-intervention (10 weeks)
  The IRO is an 85-item assessment that measures a child's level of reading participation in 17 categories (storybooks, school books, school worksheets, chalk and white boards, posters, comic books, magazines, computers, e-readers, smart phones, television shows, game consoles, board games, labels, community signs and symbols, bulletin boards, and notebooks). Using a 5-item Likert scale, the 17 categories are measured with regard to (1) five separate reading dimensions (preference, mastery, frequency, contexts an environments, social support, and available resources), (2) three physical contexts (home, school, and community), and (3) five social contexts (reading with parents, other family members, friends, classmates, and teachers). Administration requires approximately 15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Gutman, MD, Principal Investigator — Professor of Rehabilitation and Regenerative Medicine
Locations (1):
- NYC Elementary Public School (recruitment location), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bennett IM, Frasso R, Bellamy SL, Wortham S, Gross KS. Pre-teen literacy and subsequent teenage childbearing in a US population. Contraception. 2013 Apr;87(4):459-64. doi: 10.1016/j.contraception.2012.08.020. Epub 2012 Dec 11. PMID 23245352
- See also: Hernandez, D. J. (2012). Double jeopardy: How third-grade reading skills and poverty influence high school graduation. — https://files.eric.ed.gov/fulltext/ED518818.pdf
- See also: National Center for Educational Statistics. (2012). Schools and staffing survey. — https://nces.ed.gov/surveys/sass/tables/sass1112_2013314_t1s_007.asp
- See also: Nation's Report Card. (2017). Data tools: State performance compared to the nation. — https://www.nationsreportcard.gov/profiles/stateprofile?chort=1&sub=RED&sj=&sfj=NP&st=AP&year=2017R3